CLINICAL TRIAL: NCT00061984
Title: Randomised Trial Of Single Agent Doxorubicin Versus Doxorubicin Plus Ifosfamide In The First Line Treatment Of Advanced Or Metastatic Soft Tissue Sarcoma
Brief Title: Doxorubicin With or Without Ifosfamide and Pegfilgrastim in Treating Patients With Locally Advanced or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-62012; EORTC-62012
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Sarcoma
Keywords: adult angiosarcoma; adult epithelioid sarcoma; adult fibrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult rhabdomyosarcoma; adult synovial sarcoma; stage III adult soft tissue sarcoma; adult malignant fibrous histiocytoma; adult neurofibrosarcoma; stage II adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma; Hemangiosarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Rhabdomyosarcoma; Sarcoma, Synovial; Histiocytoma, Malignant Fibrous; Neurofibrosarcoma | interventions — pegfilgrastim; Doxorubicin; Ifosfamide; Combined Modality Therapy

INTERVENTIONS:
Biological: pegfilgrastim
Drug: doxorubicin hydrochloride
Drug: ifosfamide
Procedure: multimodality therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as doxorubicin and ifosfamide use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors, such as pegfilgrastim, cause the body to make blood cells. It is not yet known whether doxorubicin alone is more effective with or without ifosfamide and pegfilgrastim in treating soft tissue sarcoma.

PURPOSE: This randomized phase III trial is studying giving doxorubicin alone to see how well it works compared to giving doxorubicin together with ifosfamide and pegfilgrastim in treating patients with locally advanced or metastatic soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the progression-free and overall survival of patients with locally advanced or metastatic soft tissue sarcoma treated with doxorubicin with vs without ifosfamide and pegfilgrastim as first-line therapy.
* Compare the response in patients treated with these regimens.
* Compare the treatment-related mortality of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to WHO performance status (0 vs 1), age group (less than 50 years of age vs 50 years of age and over), presence of liver metastases (yes vs no), histological grade (2 vs 3), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive doxorubicin IV on day 1 (or IV continuously on days 1-3).
* Arm II: Patients receive doxorubicin IV on days 1-3 and ifosfamide IV over 4 hours on days 1-4. Patients also receive pegfilgrastim subcutaneously on day 5.

In both arms, treatment repeats every 3 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 8 weeks until disease progression and then every 12 weeks thereafter.

PROJECTED ACCRUAL: A total of 450 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed soft tissue sarcoma

  * Locally advanced unresectable* OR metastatic disease
  * High-grade (grade 2-3) disease according to the FNLCC grading system NOTE: *Disease that could prove resectable (including pulmonary metastasectomy) after a response to chemotherapy is allowed
* The following tumor types are eligible:

  * Malignant fibrous histiocytoma
  * Myxoid and round cell liposarcoma, pleomorphic liposarcoma, or dedifferentiated liposarcoma
  * Pleomorphic rhabdomyosarcoma
  * Synovial sarcoma
  * Myxofibrosarcoma, intermediate and high-grade
  * Fibrosarcoma
  * Leiomyosarcoma
  * Angiosarcoma
  * Malignant peripheral nerve sheath tumor
  * Epithelioid sarcoma
  * Alveolar rhabdomyosarcoma
  * Unclassifiable sarcoma, not otherwise specified
* The following tumor types are not eligible:

  * Gastrointestinal stromal tumor
  * Mixed mesodermal tumor
  * Chondrosarcoma
  * Malignant mesothelioma
  * Neuroblastoma
  * Osteosarcoma
  * Ewing's sarcoma/primitive neuroectodermal tumor
  * Desmoplastic small round cell tumor
  * Embryonal rhabdomyosarcoma
  * Alveolar soft part sarcoma
* Must have a measurable lesion with clinical evidence of progression within the past 6 weeks

  * Osseous lesions and pleural effusions are not considered measurable
* No known or symptomatic CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 60

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.8 mg/dL
* Albumin at least 2.5 g/dL

Renal

* Creatinine no greater than 1.4 mg/dL OR
* Creatinine clearance greater than 65 mL/min

Cardiovascular

* No history of cardiovascular disease

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other severe medical illness
* No psychosis
* No other prior or concurrent malignancy except adequately treated carcinoma in situ of the cervix or basal cell skin cancer
* No psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up schedule

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for advanced or metastatic disease
* Prior adjuvant chemotherapy allowed provided there was no disease progression within 6 months after completion of treatment

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to the sole index lesion

Surgery

* Not specified

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 455 (Actual)
Dates: Start 2003-04; Primary Completion 2010-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Response as assessed by RECIST criteria
Toxicity as assessed by CTC 2.0
Treatment-related mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ian R. Judson, MA, MD, FRCP, Study Chair — Institute of Cancer Research, United Kingdom
Locations (41):
- Karl-Franzens-University Graz, Graz, Austria
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Canada (5):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - McGill Cancer Centre at McGill University, Montreal, Quebec
- Denmark (2):
  - Aarhus Universitetshospital - Aarhus Sygehus, Aarhus
  - Copenhagen County Herlev University Hospital, Copenhagen
- France (3):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - CHU de la Timone, Marseille
- Germany (7):
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Universitaetsklinikum Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum der Stadt Mannheim, Mannheim
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
- Netherlands (5):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - University Medical Center Rotterdam at Erasmus Medical Center, Rotterdam
- National Cancer Institute - Bratislava, Bratislava, Slovakia
- Spain (2):
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Universitario San Carlos, Madrid
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (11):
  - Queen Elizabeth Hospital at University Hospital of Birmingham NHS Trust, Birmingham, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Royal Marsden - London, London, England
  - University College of London Hospitals, London, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Derriford Hospital, Plymouth, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Western Infirmary, Glasgow, Scotland
  - Gartnavel General Hospital, Glasgow, Scotland

REFERENCES:
- [Derived] Judson I, Verweij J, Gelderblom H, Hartmann JT, Schoffski P, Blay JY, Kerst JM, Sufliarsky J, Whelan J, Hohenberger P, Krarup-Hansen A, Alcindor T, Marreaud S, Litiere S, Hermans C, Fisher C, Hogendoorn PC, dei Tos AP, van der Graaf WT; European Organisation and Treatment of Cancer Soft Tissue and Bone Sarcoma Group. Doxorubicin alone versus intensified doxorubicin plus ifosfamide for first-line treatment of advanced or metastatic soft-tissue sarcoma: a randomised controlled phase 3 trial. Lancet Oncol. 2014 Apr;15(4):415-23. doi: 10.1016/S1470-2045(14)70063-4. Epub 2014 Mar 5. PMID 24618336